CLINICAL TRIAL: NCT06984913
Title: Ultrasound-Guided Versus Brainlab Navigation Sphenopalatine Ganglion Block in Functional Endoscopic Sinus Surgery: A Randomized Clinical Trial
Brief Title: Ultrasound-Guided Versus Brainlab Navigation Sphenopalatine Ganglion Block in Functional Endoscopic Sinus Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mostafa Ismail Sharaf, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36264PR1183/4/25
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Ultrasound; Brainlab Navigation; Sphenopalatine Ganglion Block; Functional Endoscopic Sinus Surgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ultrasound group (Experimental): Patients will receive an ultrasound-guided sphenopalatine ganglion block (4 ml bupivacaine 0.25%).
  Interventions: Other: Ultrasound-guided sphenopalatine ganglion block
- Brainlab group (Experimental): Patients will receive a Brainlab navigation sphenopalatine ganglion block (4 ml bupivacaine 0.25%).
  Interventions: Other: Brainlab navigation sphenopalatine ganglion block
- Low dose Brainlab group (Experimental): Patients will receive a Brainlab navigation sphenopalatine ganglion block (2 ml bupivacaine 0.25%) (low dose).
  Interventions: Other: Low dose Brainlab navigation sphenopalatine ganglion block

INTERVENTIONS:
Other: Ultrasound-guided sphenopalatine ganglion block — Patients will receive an ultrasound-guided sphenopalatine ganglion block (4 ml bupivacaine 0.25%).
  Arms: Ultrasound group
Other: Brainlab navigation sphenopalatine ganglion block — Patients will receive a Brainlab navigation sphenopalatine ganglion block (4 ml bupivacaine 0.25%).
  Arms: Brainlab group
Other: Low dose Brainlab navigation sphenopalatine ganglion block — Patients will receive a Brainlab navigation sphenopalatine ganglion block (2 ml bupivacaine 0.25%) (low dose).
  Arms: Low dose Brainlab group

SUMMARY:
This study compares ultrasound-guided and Brainlab navigation sphenopalatine ganglion block (SPGB) in functional endoscopic sinus surgery (FESS).

DETAILED DESCRIPTION:
Functional endoscopic sinus surgery (FESS) is the treatment modality of choice for the inflammatory disease of paranasal sinuses.

Sphenopalatine ganglion block (SPGB) is a regional analgesic technique that can be used as an alternative approach to reduce blood loss and improve the operative field during FESS without the need for hypotensive agents.

Ultrasound (US)-guided nerve block is a well-established technique in regional anesthesia and offers the advantage of real-time visualization of neural and vascular structures.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years.
* Both sexes.
* American Society of Anesthesiologists (ASA) physical status I-II.
* Patients undergoing functional endoscopic sinus surgery under general anesthesia.

Exclusion Criteria:

* Patients having a history of severe renal, hepatic, respiratory, cardiac disease, or a neurological condition.
* Drug or alcohol abuse.
* Chronic pain requires major analgesics, sedatives, or corticosteroids.
* Pregnant and lactating women.
* Hypersensitivity to local anesthetic agents.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-05-22 (Actual); Primary Completion 2025-10-16 (Actual); Study Completion 2025-10-16 (Actual)

PRIMARY OUTCOMES:
Surgical field condition | 135 min post-procedure
  The Fromme-Boezaart scale (6-point scale) will be used to assess the endoscopic surgical field condition after GA induction, at the entrance of the endoscope, and after 15, 30, 45, 60, 75, 90, 105, 120, and 135 min.
  0=No bleeding (cadaveric conditions).
  1. Slight bleeding, no suctioning required.
  2. Slight bleeding, occasional suctioning required.
  3. Slight bleeding, frequent suctioning required; bleeding threatens the surgical field a few seconds after suction is removed.
  4. Moderate bleeding, frequent suctioning required, and bleeding threatens the surgical field directly after suction is removed.
  5. Severe bleeding, constant suctioning required; bleeding appears faster than can be removed by suction; surgical field severely threatened, and surgery usually not possible.

SECONDARY OUTCOMES:
Mean arterial pressure | 135 min post-procedure
  Mean arterial pressure will be recorded after induction of general anesthesia, at entrance of endoscope, after 15, 30, 45, 60, 75, 90, 105, 120, and 135 min.
Heart rate | 135 min post-procedure
  Heart rate will be recorded after induction of general anesthesia, at the entrance of the endoscope, after 15, 30, 45, 60, 75, 90, 105, 120, and 135 min.
Intraoperative fentanyl consumption | Intraoperatively
  To improve the conditions of the surgical field, hemodynamics will be managed (A fixed target of mean blood pressure around 65 mmHg should be obtained) using these medications in the following order fentanyl 0.5 ug/kg.
Intraoperative nitroglycerine consumption | Intraoperatively
  Intraoperative requirements of nitroglycerine will be calculated.
Degree of pain | 24 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the visual analogue scale (VAS). VAS (0 represents "no pain" while 10 represents "the worst pain imaginable"). VAS: will be assessed at 0, 4, 8, 12, and 24 h postoperatively
Time to extubation | One hour postoperatively
  Time to extubation: the time from discontinuing anesthesia to fulfilling extubation criteria will be recorded.
Recovery time | One hour postoperatively
  Recovery time: the time from extubation, till patients attain an Aldrete score >9, will be recorded.
Incidence of adverse events | 24 hours postoperatively
  Incidence of adverse events such as bradycardia, hypotension, nausea, vomiting, respiratory depression, or any other complication

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.